CLINICAL TRIAL: NCT00504647
Title: Diastolic Ventricular Interaction and the Effects Of Biventricular Pacing in Hypertrophic Cardiomyopathy
Brief Title: Biventricular Pacing in Hypertrophic Cardiomyopathy
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital Birmingham (Other)
Collaborators: British Heart Foundation (Other); Medtronic (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 05/Q2707/352
Record Dates: First submitted 2007-07-18; First posted 2007-07-20 (Estimated); Last update posted 2007-07-20 (Estimated); Status verified 2007-07

CONDITIONS: Hypertrophic Cardiomyopathy
Keywords: Hypertrophic; Cardiomyopathy; Diastolic; Ventricular; Interaction; Biventricular; Pacemaker
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic; Hypertrophy; Cardiomyopathies; Heart Murmurs | interventions — Cardiac Resynchronization Therapy Devices

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Biventricular Pacemaker

SUMMARY:
Hypertrophic Cardiomyopathy is an inherited condition characterized by thickening (hypertrophy) of the heart muscle. Many patients who have this condition have a reduced ability to exercise because of breatlessness, which can in some cases be severe. This appears in most cases to be due to an impairment of the filling of the heart, especially on exercise this limits the amount of blood the heart is able to pump. Several factors may contribute to this slow filling of the heart, including (1) The heart contracts and relaxes in an incoordinate way (called 'dyssynchrony') which is inefficient, and (2) The filling of the main pumping chamber (the left ventricle) may be impeded by high pressure in the other ventricle(the right ventricle)- in other words the left ventricle is 'squashed' by the right ventricle. This is known as diastolic ventricular interaction.

Although drugs can improve the filling of the heart and relieve symptoms, some patients remain very symptomatic despite these drugs.

The mechanisms responsible for the filling abnormality in patients with Hypertrophic Cardiomyopathy are similar to those seen in the much more common condition known as Heart Failure. A special type of pacemaker technique called 'Biventricular Pacing' has been shown to markedly improve symtoms in patients with heart failure. This form of pacing has been shown to improve both 'dyssynchrony' ( incoordination) and 'ventricular interaction' (squashed left heart) in patients with Heart Failure.

We propose that Biventricular pacing may similarly improve these abnormalities in patients with Hypertrophic Cardiomyopathy, resulting in an improvement of symptoms. The study will focus on patients with the condition who have severe symtoms despite being on optimal currently available drug therapy.

DETAILED DESCRIPTION:
SUBJECTS Forty Participants, who fufil the entry criteria, will be selected. These Participants will be recruited from Cardiomyopathy clinics run at two sites. These are the Cardiomyopathy Clinics at the Heart Hospital, University College London, and from the Queen Elizabeth Hospital, Birmingham.

CONSENT Written informed consent will be obtained from all participants.

CLINICAL ASSESSMENT

A History will be taken and a Clinical Examination will be carried out. A validated Quality of life questionaire will be completed ( Minnesota Living with Heart Failure).

Maximal Cardiopulmonary exercise testing will be performed on a treadmill, with breath by breath respiratory gas sampling, using a face mask.

A 12 lead ECG will be obtained. 48hr Ambulatory Heart Rhythm Monitoring

CARDIAC ULTRASOUND SCAN ASSESSMENT

To assess the function of the Heart during its contraction and filling phases, including the degree of incoordination of the Heart muscle.

PACEMAKER IMPLANTATION

A pacemaker capable of Biventricular pacing will be implanted, using a standard established technique at one of three sites ( The Heart Hospital London, St Peters Hospital Chertsey, or Queen Elizabeth Hospital Birmingham ).

24hr POST PACEMAKER IMPLANT. Assessment of mechanical dyssynchrony will be made using Ultrasound techniques which will include 2D/ M mode Echocardiography, Doppler studies, and Tissue doppler imaging. This assessment will be made with the Pacemaker off, and in Left and Right heart pacing mode.

HAEMODYNAMIC STUDIES

These will be carried out approximately two weeks following pacemaker implantation.

The test will involve Nuclear Heart Scans (Gated Equilibrium Radionuclide Ventriculography) and Acute Volume Unloading of the right and left heart chambers.

This will be carried out at the University Of Birmingham, Department of Cardiovascular Sciences We shall apply these techniques while the heart is paced in four different modes.

The nuclear heart scan is a method by which we can measure the volume of the left heart chamber. The study will involve the placement of small needle into a vein of the patients forearm. Through this we will inject a primer which will make participants red blood cells very sticky. After twenty minutes we will take a blood sample from the same needle. This sample of blood will be mixed with a radioactive tracer. The tracer will be re-injected through the same needle into the participants' vein. This tracer will allow us to measure the amount of blood inside the chambers of the participants' heart with a special camera, a gamma camera. The pictures will be taken with the participants lying on a bed throughout.

The bed we will ask participants to lie on is called a Lower Body Negative Pressure Bed. When lying on this bed the participants' legs will be inside a see through plastic dome. A belt will be placed around the participants' waist in order to create an airtight seal around their legs. The bed is attached to a vacuum that allows us to create a low pressure environment around participants' legs. This causes blood to pool inside the veins of participants' legs. This leads to Acute Volume unloading of the right and left heart chambers.

Once participants have received the injection of the radioactive tracer and are lying comfortably in the Lower Body Negative Pressure Bed we will then take measurements of the amount of blood in the participants' heart. We shall do this using the special camera.

We shall take measurements with the pacemaker in its four different pacemaker modes, and then repeat these measurements but this time with a low pressure environment produced around participants' legs in order to reduce the pressure on your heart. The test is painless apart from mild discomfort from placing one needle at the beginning. The whole test will take between one and one and half hours.

The method of administration has been performed safely by our team for a number of years now.

After a 1 hour break the Participants will do Exercise component of the Nuclear Heart Scan. This component of the study will involve no further doses of radiation, and no new needles.

Participants will be asked to lie, semi-erect, on an exercise bed for up to 90 minutes. The exercise will be in the form of a pedal bike. The pacemaker will be programmed into four different modes of heart pacing. Whilst in each mode participants will be asked to exercise to three different stages of exercise. Each stage will last 4 minutes. The levels of difficulty will be worked out from a treadmill exercise test completed by the participants prior to the pacemaker implantation. Participants will be allowed to rest between each stage of exercise. If participants complete the whole study they will have cycled for a total of 48 minutes. During each stage 4ml of blood will be taken from the needle that will have been placed in a vein during the earlier part of the study.

During each stage of exercise an image of the heart will be taken with the gamma camera, as done earlier in the study.

From these measurements we will be able to calculate the effect of the different pacing modes on the ability of the heart to pump blood on exercise.

Participants are free to stop the exercise at any time they feel they cannot continue.

RANDOMISATION AND FOLLOW UP. Following pacemaker implant, pressure studies, and Ultrasound assessment, participants will be randomized in a double blind fashion to have their pacemaker programmed to either one of the following (1) Pacemaker Off mode, ( 2 ) Left and Right Heart chamber pacemaker mode. The Participants will be paced in that specific mode for four months before repeat Clinical and Cardiac Ultrasound assessments. The mode of pacing will then be changed, and maintained for a further four months, before repeat Clinical and Ultrasound assessment. The pacing mode will be randomly selected, but no pacing mode will be repeated in any one participant. The participant and the member of the research team performing the Clinical and Ultrasound assessment of the participant, shall be blinded to the pacemaker mode.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Hypertrophic Cardiomyopathy
* Ability to perform peak exercise oxygen consumption test.

Exclusion Criteria:

* Left ventricular outflow tract gradient more than 30mmHg
* Peak Oxygen consumption more than 75% of maximum predicted.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2006-06; Study Completion 2008-08 (Estimated)

PRIMARY OUTCOMES:
Peak Exercise Oxygen Consumption. | 4 month

SECONDARY OUTCOMES:
Myocardial Asynchrony Index | 4 months
Minnesota Quality of Life Questionnaire | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael P Frenneaux, MBBS(Hons), Principal Investigator — University of Birmingham
Locations (3):
- United Kingdom (3):
  - The Queen Elizabeth, University Hospital Birmingham, Birmingham
  - University Hospital of Wales, Cardiff
  - The Heart Hospital, London

REFERENCES:
- [Derived] Ahmed I, Loudon BL, Abozguia K, Cameron D, Shivu GN, Phan TT, Maher A, Stegemann B, Chow A, Marshall H, Nightingale P, Leyva F, Vassiliou VS, McKenna WJ, Elliott P, Frenneaux MP. Biventricular pacemaker therapy improves exercise capacity in patients with non-obstructive hypertrophic cardiomyopathy via augmented diastolic filling on exercise. Eur J Heart Fail. 2020 Jul;22(7):1263-1272. doi: 10.1002/ejhf.1722. Epub 2020 Jan 23. PMID 31975494